CLINICAL TRIAL: NCT05646069
Title: Evaluation of Novel Disposable Flexible Ureteroscope for the Treatment of Renal Calculi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Professor of Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00217933
Record Dates: First submitted 2022-11-18; First posted 2022-12-12 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: UTI; Stone, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Storz Flex-XC1 disposable flexible ureteroscope (Experimental): A patient is randomized to the experimental arm using the Storz Flex-XC1 disposable flexible ureteroscope.
  Interventions: Device: Storz Flex-XC1 Disposable Flexible Ureteroscope
- Analogue scope (No Intervention): A patient is not randomized to the experimental arm using the Storz Flex-XC1 disposable flexible ureteroscope.
- Digital ureteroscope (Experimental): A patient is randomized to the experimental arm using a Digital ureteroscope.
  Interventions: Device: Storz Flexible Digital Ureteroscope

INTERVENTIONS:
Device: Storz Flex-XC1 Disposable Flexible Ureteroscope — Patients will receive flexible ureteroscopy with the Storz Flex-XC1 disposable flexible ureteroscope.
  Arms: Storz Flex-XC1 disposable flexible ureteroscope
Device: Storz Flexible Digital Ureteroscope — Patients will receive flexible ureteroscopy with the Storz flexible Digital ureteroscope.
  Arms: Digital ureteroscope

SUMMARY:
This study is designed to provide an evaluation of currently available disposable flexible ureteroscopes in real-world conditions. Due to high re-processing costs associated with re-usable flexible ureteroscopes, there has been a demand for Urologic device manufacturers to provide single-use flexible ureteroscopes.

DETAILED DESCRIPTION:
Patients randomized to the experimental group will receive flexible ureteroscopy with the Storz Flex-XC1 disposable flexible ureteroscope.

Data will be collected and stored electronically in REDCap. Quality assurance steps will include testing of the database, including any potential data calculated by command functions within REDCap

Scope performance survey will be administered with REDcap.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18-89 undergoing ureteroscopy for laser treatment of renal calculi
* Willing to sign the Informed Consent Form
* Able to read, understand, and complete patient questionnaires, pain texts, and medication diary.

Exclusion Criteria:

* Patients having a concomitant procedure along with ureteroscopy (example: contralateral PCNL)
* Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Scope performance | 0-1 day
  Difference in scope performance grading by multiple blinded reviewers

SECONDARY OUTCOMES:
Operating room outcomes | 0-1 day
  The difference in operating room outcomes: basketing time
Operating room outcomes | 0-1 day
  The difference in operating room outcomes: scope setup time
Operating room outcomes | 0-1 day
  The difference in operating room outcomes: laser-use time
Operating room outcomes | 0-1 day
  The difference in operating room outcomes: operative time
Operating room outcomes | 0-1 day
  The difference in operating room outcomes: number of flexible ureteroscopes used
Post-operative outcomes | 4-6 weeks
  The difference in postoperative outcomes using a questionnaire: the patient has a UTI
Post-operative outcomes | 4-6 weeks
  The difference in postoperative outcomes using a questionnaire: the patient is stone-free
Post-operative surgery satisfaction of the flexible utereoscope using a questionnaire: visual quality (resolution) | 4-6 weeks
  Post-operative, the surgeon will watch videos of each surgery to analyze the satisfaction of the flexible ureteroscope (graded on a scale of 1-5)
Post-operative surgery satisfaction of the flexible utereoscope using a questionnaire: visual quality (color) | 4-6 weeks
  Post-operative, the surgeon will watch videos of each surgery to analyze the satisfaction of the flexible ureteroscope (graded on a scale of 1-5)
Post-operative surgery satisfaction of the flexible utereoscope using a questionnaire: color interference | 4-6 weeks
  Post-operative, the surgeon will watch videos of each surgery to analyze the satisfaction of the flexible ureteroscope (graded on a scale of 1-5)
Post-operative surgery satisfaction of the flexible utereoscope using a questionnaire: laser interference | 4-6 weeks
  Post-operative, the surgeon will watch videos of each surgery to analyze the satisfaction of the flexible ureteroscope (graded on a scale of 1-5)
Post-operative surgery satisfaction of the flexible utereoscope using a questionnaire: field of view | 4-6 weeks
  Post-operative, the surgeon will watch videos of each surgery to analyze the satisfaction of the flexible ureteroscope (graded on a scale of 1-5)
Post-operative surgery satisfaction of the flexible utereoscope using a questionnaire: overall impression | 4-6 weeks
  Post-operative, the surgeon will watch videos of each surgery to analyze the satisfaction of the flexible ureteroscope (graded on a scale of 1-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wong C, Xu P, Dean N, Assmus M, McDonald A, Agarwal D, Ali S, Abedi G, Margolin E, Medairos R, Nottingham C, Krambeck A. A prospective survey evaluating the visual quality of KARL STORZ fiberoptic, digital, and disposable flexible ureteroscopes. World J Urol. 2025 Feb 12;43(1):119. doi: 10.1007/s00345-025-05502-x. PMID 39937281